CLINICAL TRIAL: NCT02633696
Title: Open Label, Randomized, 2 Way-crossover Study to Investigate the Absolute Bioavailability of Oral Sylibin
Brief Title: Study to Investigate the Absolute Bioavailability of Oral Sylibin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PK-SIL-FARMA03
Record Dates: First submitted 2015-12-10; First posted 2015-12-17 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers
Keywords: Clinical trial; Phase I; Healthy volunteers; Clinical Pharmacology; Bioavailability; Silybin; Liver Trasplantation
MeSH Terms: interventions — IdB 1016

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Legalón Sil i.v 350 mg (Active Comparator): 8 healthy volunteers received 1 vial of 350 mg iv of sylibin lyophilisate for solution for infusion (legalon sil) in two hours (single dose).
  Interventions: Drug: Legalón SIL
- Silybin-phosphatidylcholine oral 360 mg (Experimental): 8 healthy volunteers received 9 capsules of 40 mg of sylibin each one (360 mg in total) orally.
  Interventions: Drug: silybin phosphatidylcholine

INTERVENTIONS:
Drug: silybin phosphatidylcholine
  Arms: Silybin-phosphatidylcholine oral 360 mg
Drug: Legalón SIL
  Arms: Legalón Sil i.v 350 mg

SUMMARY:
This clinical trial phase I in healthy volunteers is intended to describe the oral bioavailability of the silybin-phosphatidylcholine complex by calculating the area under the curve (AUC0-? and AUC0-12) after administration of the same dose of oral silybin (AUCo) and intravenous silybin (AUC iv).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals men who give their written consent to participate in the study, after having received information about the design, the project objectives, the risks and that at any moment they can refuse their cooperation.
* Understand the purpose of the study and be available for performing hospital visits and and admissions.
* Age between 18 and 45 years.
* Healthy subjects, without any organic or psychological pathology
* Clinical history and physical examination within normal limits.
* Lack of clinically relevant abnormalities in blood test (hematology, biochemistry, virology) and urine test
* Vital signs and electrocardiographic recording in the normal range.
* Males with childbearing potential partners must agree to use a highly effective method of contraception (such as surgical sterilization, double barrier method) from the moment of signing the informed consent until 6 months after the end of their participation in the study.

Exclusion Criteria:

* Subjects suffering from organic or psychological pathology. Prior to the inclusion of any volunteer it should be considered all security parameters mentioned in the protocol (biochemical markers of kidney damage and / or liver out of the normal range set by the laboratory).
* Subjects who have received prescription drug treatment in the last 15 days or any medication within 48 hours before receiving study medication.
* Subjects with a BMI that is not between 18 and 30.
* Known hypersensitivity to any drug
* Suspected of drug abuse
* Consumers of alcohol daily and / or acute alcohol poisoning in the last week.
* Subjects smoking.
* Have donated blood in the last three months.
* Participation in any other investigational drug study in the previous 3 months
* Not to be able to follow instructions or collaborate during the course of the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Sylibin pharmacokinetic parameters: Maximum plasma concentration (Cmax) obtained in the different treatment groups. | 1 Month
  Patient will be hospitalized in the clinical trial unit in order to obtain plasma concentrations previous to the administration of the corresponding dose and at the following times post-administration: : 20min, 40min, 1h, 1h20min, 1h40min 2h, 2h30min, 3h, 4h, 6h, 8h and 12h. Two more plasma concentrations will be obtained at 5 min and 10 mins post- administration of the iv dose. These measures will be calculated in order to describe the bioavailability of oral sylibinobtained in the different treatment groups.
Sylibin pharmacokinetic parameters: Area under the curve (AUC) obtained in the different treatment groups. | 1 Month
  Patient will be hospitalized in the clinical trial unit in order to obtain plasma concentrations previous to the administration of the corresponding dose and at the following times post-administration: : 20min, 40min, 1h, 1h20min, 1h40min 2h, 2h30min, 3h, 4h, 6h, 8h and 12h. Two more plasma concentrations will be obtained at 5 min and 10 mins post- administration of the iv dose. These measures will be calculated in order to describe the bioavailability of oral sylibinobtained in the different treatment groups.

SECONDARY OUTCOMES:
Sylibin pharmacokinetic parameters:Tmax, obtained in the different treatment groups. | 1 Month
Sylibin pharmacokinetic parameters:t1/2, obtained in the different treatment groups. | 1 Month
To estimate the inter and intraindividual coefficient of variation (CV) | 1 Month
To evaluate the safety (adverse events, laboratory abnormalities) and tolerability | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Aguilar, MD, Principal Investigator — Hospital Universitario Ramon y Cajal
Locations (1):
- Hospital Ramón y Cajal, Madrid, Madrid, Spain